CLINICAL TRIAL: NCT01548755
Title: Workload Assessment of a Home Monitoring Based Follow up for Biotronik ICD and CRTD Patients.
Brief Title: The Western Galilee Hospital in Nahariya Home Monitoring Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ron sela (Other Government)
Responsible Party: Sponsor-Investigator, ron sela, Ron Sela, MD, Western Galilee Hospital-Nahariya
Organization: Western Galilee Hospital-Nahariya (Other Government)
Other Study IDs: HMR_Naharia
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Tachycardia
Keywords: Home monitoring; cardiomessenger; ICD
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to study workload assessment of home monitoring based follow up for ICD or CRTD implanted patient.

DETAILED DESCRIPTION:
EP unit device clinic is a very busy clinic. Every 6 month the patients arrive for device follow up where the device parameters, patient condition and arrhythmic events are being reviewed, and reprogramming of the device (if needed) is done. Average net time of patient's stay in the clinic is between 30-45 minutes.

Patients implanted with the Lumax device family allows for a better automated follow up procedure via remote management (Home Monitoring).

The purpose of the registry is to assess workload of a Home Monitoring based follow up for Biotronik ICD and CRTD patients.

ELIGIBILITY:
Inclusion Criteria:

* Approved indication for ICD or CRTD.
* Implanted with or replaced with a Biotronik Lumax device.
* Patient is willing and able to sign consent form.
* Willing and able to attend clinic visits and follow up schedule.
* Transmission of more than 80% at 3-month FU.
* Patient older than 18 years.

Exclusion Criteria:

* No indication for ICD or CRTD implant.
* Life expectancy shorter than 12 months.
* Pregnancy.
* Participation in other clinical studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD or CRTD implanted patient
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Study Completion 2015-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Sela, MD, Principal Investigator — The Western Galilee Hospital in Nahariya
Locations (1):
- The Western Galilee Hospital in Nahariya, Nahariya, Israel